CLINICAL TRIAL: NCT01364727
Title: A Phase II Study of Amrubicin in Relapsed or Refractory Thymic Malignancies
Brief Title: A Phase 2 Study of Amrubicin in Relapsed or Refractory Thymic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heather Wakelee (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Heather Wakelee, Professor-Med, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-20444; SU-01142011-7369 (Other: Stanford University); THOR0003 (Other: OnCore)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Thymoma; Thymus Cancer; Thymic Carcinoma
MeSH Terms: conditions — Thymoma; Thymus Neoplasms | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Amrubicin (Experimental): Amrubicin 35mg/m2 IV days 1-3 every 3 weeks
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — 35 mg/m2; IV on days 1-3 each 3 week cycle
  Other Names: Calsed

SUMMARY:
A research study of the drug amrubicin in patients with cancer of the thymus (thymoma or thymic carcinoma). We hope to learn whether this drug is an effective and safe treatment for thymic cancers.

DETAILED DESCRIPTION:
Amrubicin, a synthetic 9-aminoanthracycline, is structurally similar to doxorubicin, but has a different primary mode of action. It acts primarily as an inhibitor of DNA topoisomerase II, exerting its cytotoxic effects by stabilizing a topoisomerase II mediated cleavable complex. This inhibition is significantly more than that seen in doxorubicin, which, in contrast, tends to demonstrate more DNA intercalation than amrubicin.

It has not yet been evaluated for use in thymic malignancies, but given its efficacy in NSCLC and small cell lung cancer (SCLC), as well as the known efficacy of other anthracyclines and topoisomerase II inhibitors in first-line thymoma treatment, it warrants study for use in the second line and beyond in refractory or relapsed patients. Unlike doxorubicin, amrubicin has had minimal cardiotoxicity even with ongoing use, which also makes it a promising agent for use in the second line even for patients who have previously been exposed to, and potentially helped by, doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive or metastatic thymoma or thymic carcinoma. Locally invasive disease is acceptable, provided it is not resectable.
* Previous treatment with at least one prior chemotherapy regimen.
* Documented progressive disease after the most recent chemotherapy regimen.
* Presence of measurable disease on imaging within 4 weeks prior to first dose
* Completion of prior systemic therapy at least 4 weeks prior to first dose.
* Any prior immunotherapy therapy completed at least 8 weeks prior to first dose.
* Any prior surgery completed at least 4 weeks prior to first dose, with adequate recovered from surgery.
* Any prior radiation therapy must have no residual toxic effects of therapy. Chest radiotherapy with curative intent to the primary disease complex must have been completed ≥ 28 days prior to first dose. Cranial radiation must have been completed ≥ 21 days prior to first dose. Radiotherapy to all other areas must have been completed ≥ 7 days prior to first dose.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Leukocytes ≥ 3000/mm³
* Absolute neutrophil count ≥ 1500/mm³
* Platelets ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/d
* Serum bilirubin < 1.5 x institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) and alanine transaminase (ALT) ratio < 3 x ULN
* Serum creatinine < 1.5 times institutional upper limit of normal if serum creatinine above institutional upper limit of normal, calculated serum creatinine clearance by the Cockcroft Gault method > 60 mL/min
* Left ventricular ejection fraction (LVEF) ≥ 50% by transthoracic echocardiogram (TTE) or multiple gated acquisition scan (MUGA)
* For females of childbearing potential, negative serum pregnancy test within 4 weeks of first dose.
* For males and females of childbearing potential, use of effective contraceptive methods during the study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Current use, or use within 4 weeks prior to first dose, of any other investigational agents.
* Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to amrubicin.
* Active malignancy requiring treatment other than thymic malignancy.
* Pregnant or nursing females due to unknown toxic effects of amrubicin on the developing fetus or in breast milk. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Symptomatic central nervous system metastatic disease. Patients with asymptomatic brain metastases allowed. If treated with surgical resection or radiation therapy, the patient must be stable for >= 2 weeks after completion of therapy. If the patient is on corticosteroids, the dose of corticosteroids, the dose of corticosteroids must have been stable for >= 2 weeks prior to first dose of study treatment, or be in the process of being tapered.
* Concurrent severe or uncontrolled medical disease (including but not limited to active systemic infection, diabetes, hypertension, coronary artery disease, congestive hear failure and mental illness) that in the opinion of the investigator would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Known history of seropositive human immunodeficiency virus (HIV) or use of immunosuppressive medications for other conditions that would, in the opinion of the investigator, increase the risk of serious neutropenic complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Wakelee, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Indiana University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants were fully screened for this study,and all 35 are included in Baseline Characteristics.
  However, 2 were ineligible and did not receive treatment, and so are not included in Outcomes nor Adverse Events.
Groups:
- Amrubicin: Amrubicin 35mg/m2 IV days 1-3 every 3 weeks until progression or toxicity
Period: Overall Study
Arm/Group | Amrubicin
Started | 35
Completed | 33
Not Completed | 2
Not completed — Not Eligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Amrubicin
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Histology [Count of Participants; unit: Participants]
  Thymic Carcinoma | 20
  Thymoma | 14
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Participants received amrubicin 35 mg/m2 IV days 1 to 3, every 3 weeks, until progression or toxicity.
  Tumor response rate was assessed radiographically by the Response Evaluation Criteria In Solid Tumors (RECIST), and the overall response rate (ORR) was expressed as the sum of the Complete Response (CR) rate and the Partial Response (PR) rate.
  RECIST criteria define when cancer patients improve ("respond"); stay the same ("stable"); or worsen ("progression") during treatments. The criteria presume that linear measures are an adequate substitute for 2-dimensional (2D) methods and includes 4 response categories:
  * CR = Disappearance of all target lesions
  * PR = 30% decrease in the sum of the longest diameter of target lesions
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions
  * Stable disease (SD) = Small changes that do not meet above criteria
Time Frame: 2 years
Population: Includes those participants with Complete Response (CR) plus those with Partial Response (PR).
Measure: Count of Participants; unit: Participants
Arm/Group | Amrubicin
Number analyzed (Participants) | 33
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 6
  Overall response rate (ORR) | 6

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Median Progression-free survival in patients with thymic malignancies treated with amrubicin
Time Frame: 2 years
Population: Some participants (2) continue to survive without progression, although a median and the 95% confidence interval (95% CI) for the 33 participants have been defined.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Amrubicin: Amrubicin 35mg/m2 IV days 1 to 3 every 3 weeks until progression or toxicity
Arm/Group | Amrubicin
Number analyzed (Participants) | 33
Months | 8.5 [6.7 to 38.0]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) is the sum of Complete Response (CR) rate + Partial Response (PR) rate + Stable Disease (SD) rate , and is expressed here as the sum of the Overall Response Rate (ORR = CR + PR) plus the Stable Disease (SD) rate, ORR + SD.
  Response was assessed by the RECIST criteria, elaborated above.
Time Frame: 2 years
Population: Includes those participants with Complete Response (CR) plus those with Partial Response (PR), plus those with Stable Disease).
Measure: Count of Participants; unit: Participants
Arm/Group | Amrubicin
Number analyzed (Participants) | 33
Participants
  Overall Response Rate (ORR) | 6
  Stable Disease (SD) | 23
  Disease control rate (DCR) | 29

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Amrubicin
Serious Adverse Events (participants affected / at risk) | 16/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amrubicin (N=33)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amrubicin (N=33)
Abdominal pain (General disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 5 (5)
Allergic reaction (Immune system disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 32 (32)
Anorectal infection (Infections and infestations) | 3 (3)
Anorexia (Gastrointestinal disorders) | 16 (16)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bladder infection (Infections and infestations) | 1 (1)
lymph nodes palpable (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (2)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Breast pain (General disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Buttock pain (General disorders) | 2 (2)
Cardiac disorders (Cardiac disorders) | 7 (7) — Including: Bigeminal Rhythm, chest tightness, collateral veins, mitral regurgitation, persistently split S2 and systolic murmur
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (Investigations) | 1 (1)
Conjunctivitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 18 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (27) — Including: productive
Creatinine increased (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Dizziness (General disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Edema (Blood and lymphatic system disorders) | 9 (9) — Including: Face, trunk, neck and limbs
Ejection fraction decreased (Investigations) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
eye lacrimation (Eye disorders) | 1 (1)
Fatigue (General disorders) | 33 (33)
Fever (General disorders) | 9 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Gastrointestinal disorder and pain (Gastrointestinal disorders) | 10 (10) — Including: bloody stool, Epigastric pain, esophageal spasms, perirectal abscess, rectal tenesmus and Thrush
Night sweats (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Endocrine disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Infections and infestations (Infections and infestations) | 14 (14) — Including: C.diff infection, diverticulitis, gastroenteritis, Herpes Zoster, sinus infection, Thrush and other.
Insomnia (Psychiatric disorders) | 5 (5)
Investigations (Investigations) | 5 (5) — Including: Blood CO2 elevated, blue finger, pancytopenia, white blood count increased and other
Lethargy (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 29 (29)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, left chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) — including: left chest pain and right rib pain
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (20)
Pain (General disorders) | 25 (25) — Including: Neck pain, pain in extremetynon-cardia chest pain, oral pain and pain.
Neutrophil count decreased (Investigations) | 8 (8)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (5)
Palpitations (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 12 (12)
Portal vein thrombosis (Vascular disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
bladder calcifications (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 9 (9) — including: chest pruritis, course breath sounds, decreased breath sounds, decreased breath sounds, nasal inflammation, post nasal drip, other.
right breast gynocomastia (Reproductive system and breast disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (6) — Including: blood blister, folliculitis, mall skin lesion or bite and Tenia Versicolor.
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
anal exam (Surgical and medical procedures) | 1 (1)
colonoscopy (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Thromboembolic event (Blood and lymphatic system disorders) | 2 (2)
Tooth infection (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary tract infection and pain (Psychiatric disorders) | 5 (5)
White blood cell decreased (Blood and lymphatic system disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vertigo (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Voice alteration (General disorders) | 1 (1)
Vascular disorders (Cardiac disorders) | 2 (2) — Including: Prominent chest veins and Port thrombus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No